CLINICAL TRIAL: NCT01402544
Title: Clinical Assessment Of Age-related Macular Degeneration Patients After Early Diagnosis and Treatment With Ranibizumab (COMPASS)
Brief Title: Clinical Assessment Of Age-related Macular Degeneration Patients After Early Diagnosis and Treatment With Ranibizumab
Acronym: COMPASS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Per study sponsor decision.
Sponsor: University of California, San Diego (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Henry Ferreyra, Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110567
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: AMD; Choroidal neovascularization; Ranibizumab; Age-related Macular Degeneration; Genome
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab 0.5 mg (Other): Ranibizumab 0.5 mg Intravitreal Injection, monthly, open-label, for the duration of 1 year
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5mg intravitreal injection, monthly for 12 months, or until BCVA returns to pre-wet AMD baseline.
  Other Names: Lucentis

SUMMARY:
To determine if patients treated early after diagnosis of wet age-related macular degeneration can return/maintain to their baseline pre-disease BCVA.

DETAILED DESCRIPTION:
We will conduct an open label, multi-center study of naïve AMD patients that are identified early upon disease progression (had a normal VA, FA or OCT within 4 months prior to entry) to assess if treating with ranibizumab monthly can restore all patients to their baseline vision pre-AMD. Recent randomized clinical trials (MARINA, ANCHOR) have conclusively demonstrated that continued intravitreal therapy with ranibizumab in patients with subfoveal CNV from AMD leads to stabilization of vision in over 90% of patients and improvement in vision in at least a third of the patients and has led to the approval of ranibizumab (0.5 mg) for the treatment of neovascular AMD.

Patients will receive monthly intravitreal ranibizumab injections for 12 months (with dose holding for return to baseline/ 20/20 or better and no evidence of fluid on SD-OCT or FA). All patients will have ETDRS vision and SD-OCT, and complete exam at each monthly visit. Patients will each have a blood analysis for genetics (either during the GALLEY study in which they converted to wet AMD and entered COMPASS or during this study).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Naïve wet-AMD within 4 months of disease onset (for GALLEY patients) and within 3 months of disease onset for all others
* Patients that have lost > 5 letters from baseline best vision
* BCVA 20/25-20/320

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial which includes an intervention (Patients could be participating in a non-interventional study such as the GALLEY study)
* Juxtafoveal and extrafoveal wet-AMD

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ferreyra, MD, Study Chair — University of California, San Diego
Locations (4):
- United States (4):
  - California Retina Consultants, Bakersfield, California
  - Shiley Eye Center, UCSD, La Jolla, California
  - California Retina Consultants, Santa Barbara, California
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Principal Investigator is no longer affiliated with institution. All efforts were exhausted to obtain data from all sites for this study, but we only have access to data from 'UCSD' site. Data from these participants is being reported here.
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg
Started | 12
Completed | 6
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: PI is no longer affiliated with institution. All efforts were exhausted to obtain data from all sites for this study, but we only have access to data from UCSD site. Data from these participants is being reported here
Arm/Group | Ranibizumab 0.5 mg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.42 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — PI is no longer affiliated with institution. All efforts were exhausted to obtain data from all sites for this study, but we only have access to data from UCSD site. Data from these participants is being reported here
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 12
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: PI is no longer affiliated with institution. All efforts were exhausted to obtain data from all sites for this study, but we only have access to data from UCSD site. Data from these participants is being reported here
  participants
    United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Achieve Their Pre-wet Age-Related Macular Degeneration (AMD) Baseline Visual Acuity Within 12 Months
Description: PI is no longer affiliated with institution. All efforts were exhausted to obtain data from all sites for this study, but we only have access to data from UCSD site. Data from these participants is being reported here.
Time Frame: Baseline, Month 6 and Month 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.5 mg
Number analyzed (Participants) | 6
Participants | 3

2. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) From Baseline to 6 Months and Baseline to 12 Months.
Description: Mean change was measured by letters gained or lost. A positive number is letters gained, and a negative number is letters lost.
Time Frame: Baseline, Month 6 and Month 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab 0.5 mg
Number analyzed (Participants) | 6
letters
  Change from Baseline to Month 6 | -3.333 (4.082)
  Change from Baseline to Month 12 | -9.167 (9.174)

3. Secondary Outcome: Mean Change in Central Foveal Thickness (CFT) From Baseline to 6 Months and Baseline to 12 Months
Time Frame: Baseline, Month 6 and Month 12
Population: PI is no longer affiliated with institution. All efforts were exhausted to obtain data from all sites for this study, but we only have access to data from UCSD site. Data from these participants is being reported here.The CFT image for one participant could not be located, so only 5 of the 6 enrolled participants data are being reported.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Ranibizumab 0.5 mg
Number analyzed (Participants) | 5
microns
  Change from Baseline to Month 6 | -23.4 (25.126)
  Change from Baseline to Month 12 | -25.2 (21.029)

ADVERSE EVENTS:
Description: PI is no longer affiliated with institution. All efforts were exhausted to obtain data from all sites for this study, but we only have access to data from UCSD site. Data from these participants is being reported here
Arm/Group | Ranibizumab 0.5 mg
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab 0.5 mg (N=12)
Non-ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Decrease/Blurry Vision (Eye disorders) | 1 (1)
Eye Pain (Eye disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes